CLINICAL TRIAL: NCT02647593
Title: The Clinical Characteristics of the Patients With Choledocholithiasis Without Cholangitis Showing the High Level of Aminotransferase and the Establishment of New Nomenclature ; Gallstone Hepatitis
Brief Title: The Clinical Characteristics of the Patients With Choledocholithiasis Without Cholangitis
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Dong Ki Lee, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2012-0165
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- gallstone hepatitis group,: gallstone hepatitis group (Among patients diagnosed as CBD stone who displayed above 400 IU/L of aminotransferase without cholangitis),
- control group: control group (Among patients diagnosed as CBD stone who showed the normal value of aminotransferase)

SUMMARY:
Laboratory change induced by common bile duct (CBD) stone is in general observed as the higher elevation of alkaline phosphatase (ALP) and gamma-glutamyl transpeptideas (ɤ-GT), in comparison to those of aspartate aminotransferase (AST) and alanine aminotransferase (ALT). However, some patients with CBD stone show the marked increased level of aminotransferase, which sometimes leads to misdiagnose those as liver disease caused by viral hepatitis, ischemia, and drug toxicity. The aim of this study is to investigate the clinicopathologic features of patients with CBD stones with the high level of aminotransferase in serum.

ELIGIBILITY:
Inclusion Criteria:

1. patients were diagnosed with CBD stone under endoscopic retrograde cholangiopancreatography (ERCP)
2. patients showing above 400 IU/L of aminotransferase when at the first admitted into hospital and the control groups is the patients displaying normal AST and ALT.

Exclusion Criteria:

* 1. underlying hepatobiliary disease 2. alcoholics 3. cholangitis

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "Patients have been diagnosed as CBD stone under endoscopic retrograde cholangiopancreatography (ERCP). Among patients, patients who displayed above 400 IU/L of aminotransferase without cholangitis (gallstone hepatitis group) and patients who showed the normal value of aminotransferase (control group) were enrolled in this study. We estimated two groups by comparing clinical features, lab finding, radiologic images, and findings under ERCP such as CBD diameter, CBD stone diameter, CBD stone number, periampullary diverticulum.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-10-02 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-01 (Actual)

PRIMARY OUTCOMES:
clinicopathologic features of patients with CBD stones with the high level of aminotransferase | 1year
  lab finding, radiologic images, and findings under ERCP such as CBD diameter, CBD stone diameter, CBD stone number, periampullary diverticulum.

IPD SHARING:
Plan to Share IPD: No